CLINICAL TRIAL: NCT06459258
Title: Throwing Velocity and Patient Reported Outcomes in Elite Level Handball Players After Completion of Shoulder-Pacemaker Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sportorthopädie Zentrum in Wien Hietzing (Other)
Collaborators: Austrian Research Group for Regenerative and Orthopedic Medicine (Other)
Responsible Party: Principal Investigator, Sebastian Rilk, MD, Sportorthopädie Zentrum in Wien Hietzing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EK22-201-1022; EK22-201-1022 (Other: Ethics Committee Vienna)
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Shoulder Dislocation
Keywords: Motion-Triggered Neuromuscular Electrical Stimulation-Enhanced Strength Training
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study group allocation is performed in a randomized and examiner-blinded fashion.
  All study authors and examiners are blinded to the group allocation until completion of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-NMES control group (Active Comparator): Subjects of the control group undergo a conventional standardized strength training program (3x/week, 30 minutes for 6 weeks) with concentric, eccentric, and functional training exercises.
  Interventions: Other: Non-Motion-triggered NMES training protocol
- NMES group (Experimental): Experimental group subjects undergo a motion-triggered NMES shoulder strengthening training program (3x/week, 30 minutes for 6 weeks) using the Shoulder Pacemaker (NCS Lab Srl, Modena, Italy), a motion activated stimulation device to strengthen muscular disbalances. This is accomplished through varying neuromuscular electrical stimulation intensity based on the angle of motion of the arm producing subtetanic contraction and provoking supraspinal neural adaptations.
  Electrode placement: electrode 1, inferior to the scapular spine (infraspinatus, teres minor, + posterior deltoid); electrode 2, medial to the medial scapula border (lower trapezius + rhomboids) .
  Sets x repetitions: 3x20; Levels: Level 1-3; Exercise 1: L1: Supported row, L2: Front raises in 45°, L3 Front raises (thumbs up); Exercise 2: L1: Resisted front raises, L2: Crossbody resisted raises, L3: Crossbody 'forehand swing'; Exercise 3: L1: Rear dealt fly, L2: Single arm resisted row, L3: Underhand serve
  Interventions: Other: Motion-triggered NMES training protocol

INTERVENTIONS:
Other: Motion-triggered NMES training protocol — Experimental group subjects undergo a motion-triggered NMES shoulder strengthening training program (3x/week, 30 minutes for 6 weeks) using the Shoulder Pacemaker (NCS Lab Srl, Modena, Italy), a motion activated stimulation device to strengthen muscular disbalances. This is accomplished through varying neuromuscular electrical stimulation intensity based on the angle of motion of the arm producing subtetanic contraction and provoking supraspinal neural adaptations. Electrode placement: electrode 1, inferior to the scapular spine (infraspinatus, teres minor, + posterior deltoid); electrode 2, medial to the medial scapula border (lower trapezius + rhomboids) . Sets x repetitions: 3x20 Levels: Level 1-3; Exercise 1: L1: Supported row, L2: Front raises in 45°, L3 Front raises (thumbs up) Exercise 2: L1: Resisted front raises, L2: Crossbody resisted raises, L3: Crossbody; forehand swing; Exercise 3: L1: Rear dealt fly, L2: Single arm resisted row, L3: Underhand volleyball
  Arms: NMES group
Other: Non-Motion-triggered NMES training protocol — Arm Description: Subjects of the control group undergo a conventional standardized strength training program (3x/week, 30 minutes for 6 weeks) with concentric, eccentric, and functional training exercises.
  Arms: Non-NMES control group

SUMMARY:
The successful application of treatment protocols using motion-triggered neuromuscular electrical stimulation (NMES) for treatment-resistant functional posterior shoulder instability was recently demonstrated. The purpose of this study is to evaluate the concept of a motion-triggered NMES training protocol through objective clinical outcome parameters and its impact on external rotational (ER) shoulder strength and throwing velocity in healthy, elite-level handball players.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the concept of a motion-triggered NMES training protocol through objective clinical outcome parameters and its impact on external rotational (ER) shoulder strength and throwing velocity in healthy, elite-level handball players. It is hypothesized that a 6-week motion-triggered NMES shoulder strengthening training protocol in elite-level handball players would lead to an increase in throwing velocity due to an improved motor ability and ER shoulder strength.

ELIGIBILITY:
Inclusion Criteria:

* Elite level handball players healthy and actively competing at the time of the study
* Patients must be at least 18 years at the time of signing the informed consent
* Pregnancy must be ruled out in the case of female participants (e.g., pregnancy test)
* Patient must be available for all specified assessments throughout the study duration
* All patients are required to give written informed consent before enrollment

Exclusion Criteria:

* age <18,
* history of type I or II shoulder instability according to the Stanmore classification12,
* existing pain syndrome (defined by pain at rest or during motion that is not caused by dislocation and impedes training),
* recent shoulder surgery (<1 year).
* Contraindication to SPM treatment (e.g., cardiac pacemaker)
* Neurological disorders or nerve injuries causing the instability
* Uncontrolled alcohol or substance abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Throwing velocity (km*h-1) | Baseline to 6-week post-intervention follow-up.
  the difference in throwing velocity (km*h-1) from baseline to 6-week post-intervention follow-up.

SECONDARY OUTCOMES:
Isometric hand-held dynamometer (HHD) ER and internal rotation (IR) maximal shoulder strength | Baseline to 6-week post-intervention follow-up
  Secondary outcome was the difference in isometric hand-held dynamometer (HHD) ER and internal rotation (IR) maximal shoulder strength at final follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sportorthopädie Zentrum, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moroder P, Karpinski K, Akgun D, Danzinger V, Gerhardt C, Patzer T, Tauber M, Wellmann M, Scheibel M, Boileau P, Lambert S, Porcellini G, Audige L. Neuromuscular Electrical Stimulation-Enhanced Physical Therapist Intervention for Functional Posterior Shoulder Instability (Type B1): A Multicenter Randomized Controlled Trial. Phys Ther. 2024 Jan 1;104(1):pzad145. doi: 10.1093/ptj/pzad145. PMID 37870503
- [Result] Moroder P, Danzinger V, Maziak N, Plachel F, Pauly S, Scheibel M, Minkus M. Characteristics of functional shoulder instability. J Shoulder Elbow Surg. 2020 Jan;29(1):68-78. doi: 10.1016/j.jse.2019.05.025. Epub 2019 Aug 1. PMID 31378683
- [Result] Moroder P, Plachel F, Van-Vliet H, Adamczewski C, Danzinger V. Shoulder-Pacemaker Treatment Concept for Posterior Positional Functional Shoulder Instability: A Prospective Clinical Trial. Am J Sports Med. 2020 Jul;48(9):2097-2104. doi: 10.1177/0363546520933841. PMID 32667266